CLINICAL TRIAL: NCT02455128
Title: The Influence of Therapeutic Listening on Anxiety and Fear Related to Surgery in Patients Preoperatively of Colorectal Surgery: a Randomized Clinical Trial
Brief Title: Therapeutic Listening in Patients With Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Cláudia Mesquita, Nurse - PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACM 2015
Record Dates: First submitted 2015-05-16; First posted 2015-05-27 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Anxiety; Fear
Keywords: Anxiety; Fear; Colorectal Surgery; Colorectal Neoplasms
MeSH Terms: conditions — Anxiety Disorders; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): This group will receive the therapeutic listening.
  Interventions: Other: Therapeutic listening
- Control Group (No Intervention): This group will receive usual care offered by the hospital where the study will be conducted.

INTERVENTIONS:
Other: Therapeutic listening — Method of responding to others in order to encourage better communication and clearer understanding of personal concerns.
  Arms: Experimental Group

SUMMARY:
This is a randomized clinical trial that aims to investigate the effect of therapeutic listening anxiety and preoperative fear of patients hospitalized for surgical treatment of colorectal cancer. Physiological variables will be evaluated (heart rate, blood pressure and respiratory rate), cortisol and salivary amylase and anxiety scores by State-Trait Anxiety Inventory and fear for Surgery Fear Questionnaire. The data of the variables will be compared at two different times (before and after the intervention).

DETAILED DESCRIPTION:
To calculate the sample size was chosen when using numerical scale IDATE. Considering that you want to detect a difference of 10 points (δ) in the range with a significance level of 5% (Z1-α = 1.96), a power of 80% (Z1-β = 1.96). The result obtained was 25 subjects for each group. Information related to variances of control and intervention groups were obtained through the pilot study and a correlation of 0.5 was assumed.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age;
* be hospitalized for performing surgical oncology;
* not be performing another treatment for cancer;
* not be participating in another study;
* be clinically well and / or stable (have score less than or equal to 3 by the Eastern Cooperative Oncology Group - Performance Status).

Exclusion Criteria:

* being illiterate, a condition that will prevent the participant to answer the questionnaires and instruments of the study, which are self-administered;
* be in possession of psychiatric disorders;
* be using medication containing corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Patients will be followed on three occasions during the preoperative period, an average of 24 hours before surgery.
  Change in STAI, a questionnaire to assess anxiety levels.

SECONDARY OUTCOMES:
Blood pressure | Patients will be followed on two occasions during the preoperative period, an average of 24 hours before surgery.
  Change in Blood Pressure (Systolic and diastolic) (Unit: mmHg).
Heart rate | Patients will be followed on two occasions during the preoperative period, an average of 24 hours before surgery.
  Change in radial pulse (Unit: bpm).
Respiratory rate | Patients will be followed on two occasions during the preoperative period, an average of 24 hours before surgery.
  Change in thoracic breathing movements (Unit: bpm).
Salivary cortisol | Patients will be followed on four occasions during the preoperative period, an average of 24 hours before surgery.
  Change in salivary cortisol levels. For the collection of saliva was used Salivette Tube, cotton swab to determine cortisol (Unit: μg/dL).
Salivary amylase | Patients will be followed on two occasions during the preoperative period, an average of 24 hours before surgery.
  Change in salivary amylase levels. The system for the collection and analysis of salivary amylase comprises a disposable test strip and a portable analyzer, the Cocoro Meter (Unit: KU/L).
Surgical Fear Questionnaire (SFQ) | Patients will be followed on two occasions during the preoperative period, an average of 24 hours before surgery.
  Change in SFQ, a questionnaire to assess the levels of fear of surgery.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia ACM, Simao-Miranda TP, Carvalho AMP, Elias PCL, Pereira MDG, Carvalho EC. The effect of therapeutic listening on anxiety and fear among surgical patients: randomized controlled trial. Rev Lat Am Enfermagem. 2018 Aug 9;26:e3027. doi: 10.1590/1518-8345.2438.3027. PMID 30110103